CLINICAL TRIAL: NCT05256342
Title: Biomarkers for Prediction of Analgesic Efficacy Based on Interrelations Between Pain Modulation and EEG vs. Drugs' Mode of Action in Knee OA
Brief Title: Biomarkers for Prediction of Analgesic Efficacy in Knee OA.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 0069-21-RMB
Record Dates: First submitted 2021-05-19; First posted 2022-02-25 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Knee, Osteoarthritis (OA); Biomarkers for Prediction of OA Treatment Efficacy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Duloxetine Hydrochloride; Etoricoxib; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Duloxetine (Active Comparator): Eight weeks treatment, one pill a day. Week 1st - 30 mg a day. Weeks 2nd - 8th - 60 mg a day.
  Interventions: Drug: Duloxetine 60mg
- Etoricoxib (Active Comparator): Eight weeks treatment. 60 mg daily pill ; from the second week adding omeprazol 20 mg daily
  Interventions: Drug: Etoricoxib 60 mg; Drug: omeprazol

INTERVENTIONS:
Drug: Duloxetine 60mg — Eight weeks treatment, one pill daily.
  1st week 30mg; weeks 2-7th -- 60 mg daily.
  Other Names: Cymbalta
  Arms: Duloxetine
Drug: Etoricoxib 60 mg — One pill daily for 8 weeks
  Other Names: Arcoxia
  Arms: Etoricoxib
Drug: omeprazol — 20 mg daily; will be taken with Etoricoxib from the second week of treatment
  Other Names: Prilosec, Losec
  Arms: Etoricoxib

SUMMARY:
With high NNTs for indiscriminative use in chronic pain, treatment unavoidably entails frustrating long trial and errors. It is timely to identify biomarkers that can predict analgesic efficacy for the individual patient.

The investigators propose a framework of interrelations between patient's pain modulation profile (PMP) and the drug's mode of action (MOA) based on two principles: (1) 'fix the dysfunction', relevant for drugs whose main mode of action is to modulate central pain processing; the more the dysfunctional the better the modulating drug efficacy. For example, patients with pro-nociceptive PMP due to reduced endogenous pain inhibition, as expressed by less efficient CPM will benefit from drugs that fix this dysfunction such as SNRIs, relative to patients whose pain inhibitory capacity is well functioning. Thus, for the modulating drugs, pro-nociceptivity predicts better efficacy. (2) 'bear with the dysfunction', relevant for drugs which are mostly non-modulating, acting mainly in the periphery; the more dysfunctionalת the less the non-modulating drug efficacy. This is since efficacy is limited by the dysfunctional modulation system, despite the drug's MOA-like reduction of peripheral pain mediators. Thus, for the non-modulating drugs, for example NSAIDs, pro-nociceptivity predicts less good efficacy. The likely protocol suggests that patients with anti-nociceptive PMP should be treated primarily by non-modulating drugs, while pro-nociceptive ones should be given modulating drugs.

EEG is an additional source of relevant data on brain pain processing. Being objective and stable along time, EEG based parameters are, thus, very attractive candidates to be useful biomarkers for prediction of analgesia efficacy.

This study will focus on the patients with painful knee osteoarthritis.

The aims of this study are:

1. To identify psychophysical and neurophysiological biomarkers that can serve as predictors of response to analgesic pain modulating and non-pain modulating drugs.
2. To establish a conceptual framework of individualized pain therapy based on inter-relations between patient's parameters of pain modulation and drugs' mode of action.

DETAILED DESCRIPTION:
Study design:

The study design includes two experimental meeting sessions (before and at the end / after the treatment) which include clinical and experimental assessments. After the first experimental session, the patients will be asked to rate twice a week their daily pain along two weeks, in order to confirm their OA pain level; the patients with the mean pain score of ≥4 will be supplied with the study medications. Along the 8 weeks-long treatment period, they will provide the rating of OA pain, subjective estimation of pain alleviation and reports of side effects

Clinical assessment: Will be performed by the study physician. The data on OA severity by Kellgren and Lawrence system classification, range of motion and current OA pain (last 48 h) will be collected. In addition, all patients will fill the brief pain inventory questioner (BPI) to assess their pain characteristics. In addition, all patients will be tested for the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) for assessment of OA pain, stiffness and physical function.

Experimental session:

1. At the beginning of pre-treatment experimental session, all patients will fill a following set of psychological pain-related questioners organized in one document: (1) pain catastrophizing scale (PCS), (2) HADS anxiety and depression, (3) short-form health survey (SF-12), (5) pain sensitivity questionnaire (PSQ). In addition, basic assessment of psychomotor attention and cognitive functioning will be performed using (6) Trial making tests A and B (TMT A and B) and (7) Digits symbol substitution test (DSST). All the data will be coded and no personal data will be exposed.
2. Resting-state EEG recording. Three minutes of resting-state EEG (eyes closed) will be recorded using the 64-channel EEG recording (Brain Products GmbH, Munich, Germany).
3. Psychophysical pain assessment. All tests will be performed remotely from the painful area - on arm or hand. The following tests will be performed:

   * Electrical and mechanical temporal summation (TS). For the assessment of electrical TS, a train of 10 electrical stimuli (Digitimer DS7A, Digitimer Ltd, WelWyn Garden City, England) of 2 msec width will be delivered to the non-dominant forearm with ISI of 1 sec. Subject will rate the perceived pain after the 1st and after the 5th stimuli using verbal numerical rating scale (NRS). Mechanical TS with be assessed using ten application of 256mN dull needle (from the DFNS set for quantitative sensory assessment) aimed to evoke slight pricking sensation. The TS responses will be calculated as a difference of the perceived pain between last vs. first pain score.
   * CPM. A combination of tonic heat stimulus (up to 50oC, duration up to 20 sec; TSA, Medoc, Israel) and of 3 pressure pain threshold (PPT) measurements performed on the dominant trapezius (Algomed, Medoc, Israel; 3-sec inter-stimulus interval (ISI) will be given. Stimulus heat intensity will be individually adjusted to induce pain at intensity of 50 (on 0 - 100 numerical rating scale, NRS). These stimuli will be delivered to the dominant forearm, serving a 'test-stimulus'. After a 10 min break, the non-dominant hand will be immersed into cold water bath for a period of 60-70 sec (4-10 deg). After 10 sec of the immersion, the 'test-'stimulus' will be delivered again while the hand is still in the water. Along all stimulation period, the subjects will rate their pain perception using numerical pain scale. A CPM response will be calculated as a difference in the pain perception to the 'test-stimulus' during the immersion as compared to the 'test-stimulus' given stand-alone.

Treatment follow-up:

Phone follow-up will be performed: weekly reports at weeks 1-2 and 5-6; twice a week for weeks 3-4 and 7-8. The patients will provide their OA pain score, rating of the pain-relieving drug effect (0-100 scale) and describe the treatment-related side effects for the period of last 48 hours).

Statistical analysis

The classical statistical analysis will be based on correlations between PMP and degree of drug efficacy, represented by percentage pain reduction. We then construct 3 independent model systems, one for each of the 3 PMP parameters (CPM, TS, and EEG based connectivity). Within each model we first test the two correlations, under the presumed pain modulating and non-modulating drugs, between PMP and drug efficacy. A machine learning-based cross-validation and permutation tests will be used in order to access generalizability and statistical significance of the of the findings.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* ages 45 to 75
* radiographic representation of osteoarthritis of the knee
* minimal or moderate OA severity, based on the Kellgren and Lawrence system classification (1-3)
* knee OA pain for more than 3 months, assessed by the patients as being at level 4/10 and above on average at routine daily standing/walking activities during the last week, without medication

Exclusion Criteria:

* other more prominent pain
* previous bilateral total knee replacement (TKR) surgery
* secondary OA (post-traumatic or post-infectious, osteochondritis dissecans (OCD) and enteropathic arthritis (EA) deformity)
* significant additional health problems such as substantial painful neuropathy, diabetes above of 5 yrs, renal failure, congestive heart failure, neurological diseases that might mask the pain processing system or reduce patient's cooperation or report capabilities, and significant psychiatric disorders
* use of opioids or cannabis
* known diseases of gastrointestinal tract such as esophagitis, gastritis and duodenitis
* patients that had side effects to the study drugs in the past.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
CPM, a psychophysical parameter for pain inhibition, NPS | up to 2 years
  Post vs pre-treatment changes in Conditioned Pain Modulation (CPM)
TS, a psychophysical parameter for pain facilitation, NPS | up to 2 years
  Post vs pre-treatment changes in Temporal Summation of pain (TS)
resting-state EEG theta power, microvolts | up to 2 years
  Post vs pre-treatment changes in the EEG power within theta band
resting-state EEG alpha power, microvolts | up to 2 years
  Post vs pre-treatment changes in the EEG power within alpha band
Clincial pain, VAS | up to 2 years
  Post vs pre-treatment changes in VAS
Pain-related disability, numerical scores | up to 2 years
  Post vs pre-treatment changes (disability score)

CONTACTS AND LOCATIONS:
Overall Officials: David Yarnitsky, Prof, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No